CLINICAL TRIAL: NCT02936830
Title: Effectiveness of Nano-hydroxyapetite Care Paste in Reducing Dentinhypersenstitivity: A Double Blind Randomized Control Trial
Brief Title: Effectiveness of Nanohydroxyapetite Paste on Reducing Dentin Hypersensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Dalia Nayil Alharith, Post-graduate student, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPGRP/43533002/71
Record Dates: First submitted 2016-10-16; First posted 2016-10-18 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — sodium fluoride topical preparation; Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): 21 individuals with dentin hypersensitivity will receive a placebo solution of glycerol diluted in water in a 1:1 concentration applied on the sensitive area by the dentist
  Interventions: Drug: Glycerol
- Fluoride group (Active Comparator): 21 individuals with dentin hypersensitivity will receive 5% Sodium Fluoride varnish applied on the sensitive area by the dentist
  Interventions: Drug: 5% Sodium Fluoride Varnish
- Nanohydroxyapetite (Experimental): 21 individuals with dentin hypersensitivity will receive 15% nanohydroxyapetite paste applied on the sensitive area by the dentist
  Interventions: Drug: 15% Nanohydroxyapetite paste

INTERVENTIONS:
Drug: 5% Sodium Fluoride Varnish — 5% sodium fluoride varnish applied on the dentin by the dentist
  Other Names: Duraphat
  Arms: Fluoride group
Drug: 15% Nanohydroxyapetite paste — 15% nanohydoxyapetite paste without potassium nitrate or fluoride applied on the dentin by the dentist
  Other Names: Nanohydroxyapetite paste
  Arms: Nanohydroxyapetite
Drug: Glycerol — Glycerol with water in a 1: 1 ratio
  Other Names: glycerol water mixture
  Arms: Control

SUMMARY:
The aim of this study is to compare the efficacy of dentine hypersensitivity reduction using in office paste formula containing nanoHydroxyapatite with the commercially available fluoride (duraphat) and a placebo in treating hypersensitivity in a single visit.

DETAILED DESCRIPTION:
Following the approval of the Research Ethics Committee of Riyadh college of Dentistry and Pharmacy (The Institutional Review Board), a randomized double blind single treatment controlled clinical trial will be carried out on 60 patients (-- males and -- females) between the age group of 18 to 45 years, visiting the out-patient clinics of Riyadh Colleges of Dentistry and Pharmacy during the period between October and December.

The protocols for the study will be developed as per the guidelines for the design and conduct of clinical trials on dentinal hypersensitivity and in accordance with the Declaration of Helsinki and Guidelines for Good Clinical Practice. Prior to the start of the study patients will be given both verbal and written information about the process and an appropriate signed informed consent form will be obtained.

Only subjects demonstrating two hypersensitive teeth that satisfied the tactile and airblast hypersensitivity enrolment criteria, qualified to participate in the study. Qualified subjects will be randomly defined to one of the three study groups in order to have 20 subjects per treatment group:

* Study 1: nanoXIM care paste, fluoride-free (test group)
* Study 2: fluoride paste
* Study 3: placebo group (positive control group).

Subjects selected will undergo thorough clinical examination, followed by oral prophylaxis, oral hygiene instructions and dietary counseling. After the teeth isolation with cotton rolls, changes in the dentin sensitivity to tactile (dental explorer), thermal stimuli (drops of melted ice) and air stimuli (blast from dental syringe) will be evaluated. Following application of the stimuli, responses will be evaluated and assessed by the Visual Analog Scale (VAS). The survey form will be completed by the examiner to have a baseline prior to paste application in the first visit. The survey contains five questions, rated on a 10-point scale, assessing:

1. Degree of pain.
2. Duration of pain.
3. Intensity of pain.
4. Tolerability of pain.
5. Description of pain.

Data Analysis

The study patients will be randomly assigned into 3 groups (N, F and P) equal groups of 20. The randomization process will be made using a computer-generated random table. Excel software (Micro- soft) will be used for randomization. The pastes used on the study labeled N, F and P respectively, will be completely wrapped not allowing the pastes applicant or any other member of the research team to know what test paste will be applied on the patients. The patients will be blinded by not letting them know which agents will be applied. The chief investigator, the first author in this study, will coordinate the entire trial and recruited the various operators for the same.

ELIGIBILITY:
Inclusion Criteria:

* Hypersensitive areas on facial surfaces of the teeth (incisors, canines, premolars, and first molars with exposed cervical dentin) with at least two teeth scoring "pain (scale stimuli test, scores 2 and 3)" during application of stimulus (airblast and tactile sensitivity test)
* Good periodontal health (no probing depth > 4 mm) with no other conditions that might explain their apparent dentin hypersensitivity
* Good overall physical health
* Age between 18 and 45 years
* Provision of written informed consent
* Patient willing to participate in the study

Exclusion Criteria:

* Chipped teeth
* Defective restorations
* Fractured undisplaced canines
* Deep dental caries
* Deep periodontal pockets
* Orthodontic appliances
* Dentures or fixed dental prostheses that would interfere with the evaluation of hypersensitivity
* Periodontal surgery within the previous 6 months
* Ongoing treatment with antibiotics and/or anti- inflammatory drugs past 3 months
* Ongoing treatment for tooth hypersensitivity
* Pregnancy or lactation
* Smokers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity measured by a visual analog scale | One month
  Dentin sensitivity measured by giving the patient a visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Dalia N AlHarith, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh colleges of dentistry and pharmacy olaya campus, Riyadh, ArRiyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kunam D, Manimaran S, Sampath V, Sekar M. Evaluation of dentinal tubule occlusion and depth of penetration of nano-hydroxyapatite derived from chicken eggshell powder with and without addition of sodium fluoride: An in vitro study. J Conserv Dent. 2016 May-Jun;19(3):239-44. doi: 10.4103/0972-0707.181940. PMID 27217637
- [Background] Douglas de Oliveira DW, Oliveira ES, Mota AF, Pereira VH, Bastos VO, Gloria JC, Goncalves PF, Flecha OD. Effectiveness of Three Desensitizing Dentifrices on Cervical Dentin Hypersensitivity: A Pilot Clinical Trial. J Int Acad Periodontol. 2016 Apr 8;18(2):57-65. PMID 27128158
- [Background] Wang L, Magalhaes AC, Francisconi-Dos-Rios LF, Calabria MP, Araujo D, Buzalaf M, Lauris J, Pereira JC. Treatment of Dentin Hypersensitivity Using Nano-Hydroxyapatite Pastes: A Randomized Three-Month Clinical Trial. Oper Dent. 2016 Jul-Aug;41(4):E93-E101. doi: 10.2341/15-145-C. Epub 2016 Feb 26. PMID 26919080
- [Background] Gopinath NM, John J, Nagappan N, Prabhu S, Kumar ES. Evaluation of Dentifrice Containing Nano-hydroxyapatite for Dentinal Hypersensitivity: A Randomized Controlled Trial. J Int Oral Health. 2015 Aug;7(8):118-22. PMID 26464553